CLINICAL TRIAL: NCT01861106
Title: Allogeneic Hematopoietic Stem Cell Transplant for Patients With Mutations in GATA2 or the MonoMAC Syndrome
Brief Title: Allogeneic Hematopoietic Stem Cell Transplant for GATA2 Mutations
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130132; 13-C-0132
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2026-01-09 (Actual); Status verified 2026-01-07

CONDITIONS: GATA2; Immunodeficiency; MDS
Keywords: Allogeneic Donors; Peripheral Blood Stem Cell; Immunodeficiency; Myelodysplasia; Haploidentical
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Anemia, Refractory, with Excess of Blasts | interventions — fludarabine; fludarabine phosphate; Busulfan; Cyclophosphamide; Whole-Body Irradiation; Mycophenolic Acid; Tacrolimus; Antilymphocyte Serum

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Arm A (Active Comparator): 10/10 HLA Matched Related Donor or Unrelated Donor or 9/10 HLA with DQ mismatch Transplant
  Interventions: Procedure: Allogeneic HSCT; Drug: Busulfan Test dose; Drug: Fludarabine (Fludara, Berlex Laboratories); Drug: Busulfan (Busulfex); Drug: Mycophenolate mofetil (MMF); Drug: Tacrolimus
- Arm B (Active Comparator): 9/10 or 8/10 HLA Match Related Donor or Unrelated Donor or Haploidentical Donor Transplant
  Interventions: Procedure: Allogeneic HSCT; Drug: Busulfan Test dose; Drug: Fludarabine (Fludara, Berlex Laboratories); Drug: Busulfan (Busulfex); Drug: Cyclophosphamide (CTX, Cytoxan); Drug: Mycophenolate mofetil (MMF); Drug: Tacrolimus
- Arm C (combined with Arm B per Amendment N) (Active Comparator): Haploidentical Related Donor Transplant
  Interventions: Procedure: Allogeneic HSCT; Drug: Busulfan Test dose; Drug: Fludarabine (Fludara, Berlex Laboratories); Drug: Busulfan (Busulfex); Drug: Cyclophosphamide (CTX, Cytoxan); Procedure: Total Body Irradiation (TBI); Drug: Tacrolimus
- Arm D (Deleted this arm per amendment I) (Active Comparator): Umbilical Cord Blood Transplant
  Interventions: Procedure: Allogeneic HSCT; Drug: Fludarabine (Fludara, Berlex Laboratories); Drug: Cyclophosphamide (CTX, Cytoxan); Procedure: Total Body Irradiation (TBI); Biological: Equine Anti-Thymocyte Globulin
- Arm E (Deleted this arm per amendment O) (No Intervention): Donor

INTERVENTIONS:
Procedure: Allogeneic HSCT — Stem cell transplant
  Arms: Arm A; Arm B; Arm C (combined with Arm B per Amendment N); Arm D (Deleted this arm per amendment I)
Drug: Busulfan Test dose — 0.8 mg/kg IV infusion over 3 hours one time dose administered 5 to 14 days prior to start of preparative regimen (Days -11 to -20)
  Arms: Arm A; Arm B; Arm C (combined with Arm B per Amendment N)
Drug: Fludarabine (Fludara, Berlex Laboratories) — 40 mg/m2 IV (in the vein) over 30 minutes (in the vein) once daily on Days -6, -5, -4, and -3 or 30 mg/m2 IV over 30 minutes (in the vein) once daily on Days -6, -5, -4, -3, and -2
  Arms: Arm A; Arm B; Arm C (combined with Arm B per Amendment N); Arm D (Deleted this arm per amendment I)
Drug: Busulfan (Busulfex) — 3.2 mg/kg IV (in the vein) over 3 hours once daily on Days -6, -5, -4 and -3 (weight based dosing). If in Arm B and if poor or very poor risk clonal chromosomal abnormalities, busulfan will also be given on day -2.
  Arms: Arm A; Arm B; Arm C (combined with Arm B per Amendment N)
Drug: Cyclophosphamide (CTX, Cytoxan) — 14.5 mg/kg IV (in the vein) infusion over 30 minutes once daily on days -6 and -5 (weight based dosing) or 50 mg/kg IV infusion over 2 hours on day -6 (weight based dosing). For post-transplant, 50/kg IV once daily x2 doses on days +3 and +4
  Arms: Arm B; Arm C (combined with Arm B per Amendment N); Arm D (Deleted this arm per amendment I)
Procedure: Total Body Irradiation (TBI) — 200 cGy on Day -1
  Arms: Arm C (combined with Arm B per Amendment N); Arm D (Deleted this arm per amendment I)
Drug: Mycophenolate mofetil (MMF) — 15mg/kg IV over 2 hours BID starting on day +5 will continue until day +35 (+/- 2 days)
  Arms: Arm A; Arm B
Drug: Tacrolimus — 0.02mg/kg IV continuous infusion over 24 hours starting on day +5 until day +180
  Arms: Arm A; Arm B; Arm C (combined with Arm B per Amendment N)
Biological: Equine Anti-Thymocyte Globulin — (Deleted this intervention per amendment I): 30mg/kg IV (in the vein)once daily x 3 days on Days -6, -5, -4 (3 doses total)
  Arms: Arm D (Deleted this arm per amendment I)

SUMMARY:
Background:

- GATA2 deficiency is a disease caused by mutations in the GATA2 gene. It can cause different types of leukemia and other diseases. Researchers want to see if a stem cell transplant can be used to treat this condition. A stem cell transplant will give stem cells from a matching donor (related or unrelated) to a recipient. It will allow the donor stem cells to produce healthy bone marrow and blood cells that will attack the recipient s cancer cells.

Objectives:

- To see if stem cell transplants are successful at treating GATA2 mutations and related conditions.

Eligibility:

- Recipients who are between 6 and 70 years of age and have GATA2 deficiency.

Design:

* All participants will be screened with a physical exam and medical history. Blood samples will be collected. Recipients will have imaging studies and other tests.
* Recipients will have chemotherapy or radiation to prepare for the transplant. On the day of the transplant, they will receive the donated stem cells.
* Recipients will stay in the hospital until their condition is stable after transplant.
* Frequent blood tests and scans will be required for the first 6 months after the transplant, followed by less frequent visits over time.

DETAILED DESCRIPTION:
Background:

Genetic and sporadic mutations on one allele of the GATA2 gene lead to a syndrome termed MonoMAC. MonoMAC is characterized by: 1) infections with Mycobacterium avium complex (MAC) and other opportunistic infections, 2) deficiency of monocytes, B-lymphocytes, and Natural Killer (NK) cells in the peripheral blood, and 3) progression to myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML), and acute myelogenous leukemia (AML), and 4) mutations on one allele of GATA2 in most participants. We propose to evaluate the efficacy and safety of allogeneic hematopoietic stem cell transplantation (HSCT) using different conditioning regimens from different donor sources in reconstituting normal hematopoiesis and reversing the disease phenotype in participants with mutations in GATA2, or the clinical syndrome of MonoMAC.

Objectives: Primary:

-To determine whether allogeneic hematopoietic stem cell transplant (HSCT) approach reconstitutes normal hematopoiesis and reverses the disease phenotype by one year posttransplant in participants with mutations in GATA2 or the clinical syndrome of MonoMAC.

Eligibility:

* Recipients ages 6-70 years old with mutations in GATA2 or the clinical syndrome of MonoMAC. Clinical history of at least one serious or disfiguring infection and GATA2 bone marrow immunodeficiency disorder with loss of one or more immune populations in the bone marrow including monocytes, Natural Killer (NK) cells, and B-lymphocytes, with or without additional cytopenias involving the red blood cell, neutrophil, or platelet compartment.
* Have a 10/10 or a 9/10 or an 8/10 HLA-matched related or unrelated donor (HLA -A, -B, -C, DRB1, DQB1 by high resolution typing) or a haploidentical related donor; unrelated donors are identified through the National Marrow Donor Program.

Design: Two Arms

* Participants with mutations in GATA2, or the clinical syndrome of MonoMAC, with a 10/10 (or 9/10 matched if the mismatch is at DQ) HLA-matched related or unrelated donor will receive a pre-transplant conditioning regimen consisting of fludarabine 40 mg/m2 IV once daily for 4 days on days -6, -5, -4, and -3, busulfan based on pharmacokinetic levels from test dose or real time pharmacokinetics (PKs) (3.2 mg/kg IV will be the default dose) once daily on days -6, -5, -4, and -3, and HSCT on day 0.
* Participants with mutations in GATA2, or the clinical syndrome of MonoMAC, with a 9/10 or an 8/10 HLA-matched related or unrelated donor (if the mismatch is not at DQ) or with a haploidentical related donor, will receive a pre-transplant conditioning regimen consisting of cyclophosphamide 14.5 mg/kg IV once daily for 2 days on days -6 and -5, busulfan based on pharmacokinetic levels from test dose or real time PKs ( 3.2 mg/kg IV will be the default dose) once daily on days -4, -3, (if poor or very poor risk clonal cytogenetic abnormalities are present, then three days of busulfan IV once daily on days -4, -3, and -2 will be given), fludarabine 30 mg/m2 IV once daily for 5 days on days -6 to -2, 200 cGy TBI on day -1, and HSCT on day 0.
* Post-transplant immunosuppression for GVHD prophylaxis for recipients of all groups will consist of cyclophosphamide 50 mg/kg IV once daily for 2 days on days +3 and +4, along with mycophenolate mofetil from day +5 to approximately day +35 and tacrolimus from day +5 to approximately day +180. If there is no evidence of graft-versus- host disease, tacrolimus will be stopped or tapered at approximately day +180.

ELIGIBILITY:
* ELIGIBILITY CRITERIA:

INCLUSION CRITERIA- Recipient

1. Patient age of 6-70 years.
2. Mutation in the GATA2 gene, or evidence of loss of expression of one allele of GATA2, by cDNA analysis performed by a CLIA certified laboratory, or the clinical syndrome of MonoMAC.
3. Clinical history of at least one serious or disfiguring infection and/or GATA2 bone marrow immunodeficiency disorder with lose of one or more immune populations in the bone marrow including monocytes, Natural Killer (NK) cells, and B-lymphocytes, with or without additional cytopenias involving the red blood cell, neutrophil, or platelet compartment.
4. Availability of a 10/10 or 9/10 or 8/10 HLA-matched related or unrelated donor, or a haploidentical related donor.
5. Patients may have evidence of MDS with one or more peripheral blood cytopenias and greater than 5% blasts but must have less than 10% blasts in the bone marrow in the absence of filgrastim in order to proceed directly to transplant. The majority of patients with MDS will have less than 5% blasts.
6. Disease status: Patients are to be referred in remission for evaluation. Should a patient have progressive disease with >10% blasts on screening/baseline bone marrow biopsy, the patient may receive standard treatment under the current study prior to proceeding with transplant. Once the patient has <10% blasts, they may proceed to transplant. The patient may also be referred back to their primary hematologist or oncologist for treatment. If this course of action is not in the best interest of the patient according to the clinical judgment of the PI/LAI, then the patient may receive standard treatment for the malignant disease or hematological disorder under the current study. If under either of these settings, it becomes apparent that the participant will not be able to proceed to transplant, then he/she must come off study. Recipient-Subjects receiving a standard therapy will be told about the therapy, associated risks, benefits and alternatives of the proposed therapy, and availability of receiving the same treatment elsewhere, outside of a research protocol.
7. Left ventricular ejection fraction > 40%, preferably by 2-D echocardiogram obtained within 90 days prior to initiation of conditioning therapy.
8. Creatinine: Adult patients: <= 2.0 mg/dl and creatinine clearance >= 30 ml/min; Pediatric patients (<18 years old): creatinine <1.5 mg/dL and a creatinine clearance, using the Schwartz Formula, > 30 mL/min/1.73m^2.
9. Serum conjugated bilirubin < 2.5 mg/dl; serum ALT and AST <= 5 times upper limit of normal.
10. Pulmonary function tests: FEV1 and DLCO >30% Note: For children who are unable to cooperate for PFTs, the criterion is: No evidence of dyspnea at rest, no exercise intolerance, and no requirement for supplemental oxygen therapy
11. Ability of patient or Legally Authorized Representative (LAR) (if the patient is deemed by the treating physician to be cognitively impaired or questionably impaired in such a way that the ability of the patient to give informed consent is questionable) to understand and the willingness to sign a written informed consent document indicating that they are aware of the investigational nature of this study or written informed consent obtained from parent or legal guardian if subject is a minor.
12. As therapeutic agents used in this trial may be harmful to a fetus, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for at least one-year post-allo HSCT. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in the study, she should inform her treating physician immediately.
13. All transplant patients remain in the NIH hospital or, if discharged, stay close to the NIH for a minimum of 100 days after transplant or longer, if there are complications. An adult caregiver must be with the patient at all times from discharge to day 100.

EXCLUSION CRITERIA- Recipient

1. Patients who are receiving any other investigational agents with the exception of virus- specific cytotoxic T-cells for the treatment of viral infection/reactivation prior to allo HSCT
2. HIV-positive patients are ineligible because these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
3. History of allergic reactions attributed to compounds of similar chemical or biological composition to agents (steroids, cyclophosphamide, busulfan) used in the study
4. Chronic active hepatitis B. Patient may be hepatitis B core antibody positive. For patients with a concomitant positive hepatitis B surface antigen, patients will require a hepatology consultation. The risk-benefit profile of transplant and hepatitis B will be discussed with the patient, and eligibility determined by the PI or Lead Associate Investigator.
5. History of psychiatric disorder which may compromise compliance with transplant protocol, or which does not allow for appropriate informed consent.
6. Active infection refractory to antimicrobial therapy.
7. Active CNS involvement by malignancy (patients with known positive CSF cytology or parenchymal lesions visible by prior CT or MRI).
8. Pregnant or lactating.
9. The effects on breast-milk are unknown and may be harmful to the infant; therefore, women should not breast feed during the interval from study entry to one year post-transplant.
10. Presence of active malignancy in another organ system other than the hematopoietic, except when driven by viruses in which case the immune reconstitution after transplant may control the malignancy. This includes solid tumors not in remission.
11. No available 10/10 or 9/10 or 8/10 HLA-matched related or unrelated donor, or haploidentical related donor.

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2013-07-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine whether allogeneic HSCT approach results in engraftment and restores normal hematopoiesis by one year in patients with mutations GATA2. | 1 year after completing ASCT
  Determination that engraftment has occurred, normal hematopoiesis has been restored and the clinical phenotype after allogeneic HSCT has been reversed

SECONDARY OUTCOMES:
To determine the safety of allogeneic HSCT for patients with mutations in GATA2 | 3 years
  Fractions of patients with transplant related toxicity will be reported along with 95% confidence intervals
To determine the incidence of grade III-IV acute GVHD | 100 days
  fractions will be reported using simple estimates along with 95% two-sided confidence intervals
To determine the incidence of chronic graft-versus-host disease | 1 year and 2 years post-transplant
  Fractions of patients with transplant related toxicity as well as the fractions with aGVHD and cGVHD will be reported along with 95% confidence intervals.
To characterize the immune reconstitution inflammatory syndrome (IRIS) | Days 30, 100, 6 months, and one year post-transplant
  fraction of patients who experience a reversal of the described immunologic abnormalities will be reported along with a 95% two-sided confidence interval. Fractions will be compared using Fisher's exact test.
To characterize the immune reconstitution in 10/10 matched related and unrelated donor transplant recipients and haploidentical related donor transplants who receive GVHD prophylaxis | Days 30, 100, 6 months, and one year post-transplant
  Fractions will be compared using Fisher's exact test.
Overall survival, and disease-free survival. | 5 years post-transplant
  determined using the Kaplan-Meier method for all evaluable patients beginning at their date of transplant, along with the median value and the 95% confidence interval at the median

CONTACTS AND LOCATIONS:
Overall Officials: Danielle E Pregent-Arnold, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- [Derived] West RR, Bauer TR, Tuschong LM, Embree LJ, Calvo KR, Tillo D, Davis J, Holland SM, Hickstein DD. A novel GATA2 distal enhancer mutation results in MonoMAC syndrome in 2 second cousins. Blood Adv. 2023 Oct 24;7(20):6351-6363. doi: 10.1182/bloodadvances.2023010458. PMID 37595058
- [Derived] Wu Z, Gao S, Diamond C, Kajigaya S, Chen J, Shi R, Palmer C, Hsu AP, Calvo KR, Hickstein DD, Holland SM, Young NS. Sequencing of RNA in single cells reveals a distinct transcriptome signature of hematopoiesis in GATA2 deficiency. Blood Adv. 2020 Jun 23;4(12):2656-2670. doi: 10.1182/bloodadvances.2019001352. PMID 32556286
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2013-C-0132.html